CLINICAL TRIAL: NCT06209658
Title: The Effect of Breastfeeding Education Given to Primiparous Mothers With the Teach Back Method on Breastfeeding Self-Efficacy Perception and Anxiety Level
Brief Title: Breastfeeding Education Given to Primiparous Mothers With the Teach-Back Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, GÜLHAN AKDEMİR, teaching assistant at Igdır University, Igdir University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IgdirU
Record Dates: First submitted 2023-11-10; First posted 2024-01-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breastfeeding Self-efficacy
Keywords: teach back method; breastfeeding self-efficacy perception; anxiety level; primiparous mother; breastfeeding education

STUDY DESIGN:
Intervention Model Description: A total of 70 people, 35 in the experimental group and 35 in the control group, will be included in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): breastfeeding education with Teach Back
  Interventions: Diagnostic Test: breastfeeding education of Teach Back
- Control Group (Other): breastfeeding education simple explanation
  Interventions: Other: breastfeeding education simple explanation

INTERVENTIONS:
Diagnostic Test: breastfeeding education of Teach Back — breastfeeding education simple explanation is given and the woman is asked to explain and practice.
  Arms: experimental group
Other: breastfeeding education simple explanation — breastfeeding education simple explanation
  Arms: Control Group

SUMMARY:
The Teach-Back method was initially developed as a communication technique for patients to remember important information about their diagnosis, treatment or medication and to understand what to do. Method; It requires recalling and explaining any information learned during the interaction between the healthcare team and clients. It has been seen that the use of the tell-what-you-learned method can be used effectively in increasing the learning and comprehension level of individuals who lack health knowledge, contributing to positive health behaviors and reducing the return to health institutions, and it has begun to be used in different areas that require patient education. There are no examples of studies in which the tell-what-you-learned method, which has been brought to the agenda and implemented abroad in recent years, is used in our country.

The development of breastfeeding self-efficacy is a very challenging process. Postpartum anxiety occurs in women with low breastfeeding self-efficacy perception. Different training methods are used to initiate and maintain breastfeeding. However, there is no generally accepted method that can bridge the communication gap between patients and healthcare professionals and can be used in health education. It is important to use the tell-what-you-learned method, which is used in patient/client training and is expressed as a communication technique based on expressing what the caregivers have learned in their own words, as it is not enough for the individuals being cared for to say "I understand", in terms of increasing the success of breastfeeding and improving the health of the mother and baby.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of breastfeeding education given using the tell-what-you-learned method on breastfeeding self-efficacy perception and anxiety level.The population of the research consists of women who gave birth at Iğdır State Hospital in the last 6 months of 2022. According to the records of Iğdır Provincial Health Directorate Statistics Department, for 2022; A total of 1351 live births took place in Iğdır State Hospital in the relevant period, including 257 in July, 269 in August, 213 in September, 207 in October, 188 in November and 217 in December.

Power analysis was performed to determine the sample size. The power of the research is defined as the possibility of revealing the difference between two applications. The power of the study is expressed as 1 - ß probability of error, and in general, studies must have at least 80% power. The minimum number of individuals required to be included in the sample of the study was calculated using the G-power 3.1.9.7 program, based on the data of the study titled "The effect of antenatal education based on strengthening the perception of breastfeeding self-efficacy on the perception of breastfeeding self-efficacy and breastfeeding success". Alpha margin of error was determined as 5%, the power of the study was determined as 80% (Effect Size: 0.70), and it was observed that there should be at least 34 people in each group. A total of 68 women will be included in the sample, including 34 study and 34 control groups. Postpartum women who meet the inclusion criteria for the study will be selected to the intervention and control groups by simple randomization.Taking into account the inclusion and exclusion criteria, women will be divided into intervention and control groups by simple randomization method. A random number generation program (Research Randomizer) will be used in the randomization of the sample. The randomization process will be created by an impartial researcher who is not involved in the research. Women will not be informed about the groups they are in, only the researcher will know which group they will be in, and single blindness will be ensured in the study.Intervention and control group data in the study;

1. Personal Information Collection Form
2. Breastfeeding Self-Efficacy Scale
3. It will be collected using the Beck Anxiety Scale (BAI). The Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert-type scale consisting of 14 items (1: not at all confident and 5: always confident). The lowest score that can be obtained from the scale is 14 and the highest score is 70. A high score indicates high breastfeeding self-efficacy.Beck Anxiety Scale Beck Anxiety Scale: The lowest score that can be obtained from the scale is 0 and the highest score is 63. An increase in the score obtained from the scale indicates that the individual's anxiety increases. A total score from the scale between 8 and 15 indicates mild anxiety, between 16 and 25 indicates moderate anxiety, and between 26 and 63 indicates severe anxiety.

Research data will be evaluated using SPSS 21.0 program. Homogeneity of the groups will be evaluated by Chi Square test for categorical variables, Mann Whitney U or t test for independent groups, depending on the data for numerical variables. Multiway Analysis of Variance in Repeated Measurements will be used to compare Breastfeeding Self-Efficacy Scale mean scores in the intervention and control groups according to group, time and group-time interaction. In further analysis of the difference between the breastfeeding self-efficacy scale mean scores in the intervention and control groups, One-Way Analysis of Variance in Repeated Measurements will be used to compare the mean scores of the groups among themselves, and the T-Test in Dependent Groups with Bonferroni Correction will be used to compare the measurements with each other.

ELIGIBILITY:
Inclusion Criteria:

* Living in Iğdır city center
* Ability to read and write
* Don't be primiparous
* Giving birth at term and in a healthy manner
* Having a healthy newborn
* Having had a vaginal or cesarean birth

Exclusion Criteria:

* Living in Iğdır city center
* Ability to read and write
* Don't be primiparous
* Giving birth at term and in a healthy manner
* Having a healthy newborn
* Having had a vaginal or cesarean birth

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — giving birth for the first time
Enrollment: 70 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Collection of post-training data | two months
  Mothers will be given breastfeeding training 3 times using the Teach Back method. First breastfeeding training with teach-back method in the 2nd-5th week after birth. The second breastfeeding training takes place between days 13-17 after birth. Between days 30-42 after birth, the third breastfeeding training takes place. will be given between days. The Breastfeeding Self-Efficacy Scale will be administered after each breastfeeding training.
  The Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert-type scale consisting of 14 items (1: not at all confident and 5: always confident). The lowest score that can be obtained from the scale is 14 and the highest score is 70. A high score indicates high breastfeeding self-efficacy.
Collection of post-training data | two months
  The Beck Anxiety Scale will be administered after each breastfeeding education given with the Teach-Back method.
  The scale, consisting of 21 questions, is a 4-point Likert type. Each item in the scale is scored between 0 (not at all) and 3 (serious). The lowest score that can be obtained from the scale is 0 and the highest score is 63. An increase in the score obtained from the scale indicates that the individual's anxiety increases. A total score from the scale between 8 and 15 indicates mild anxiety, between 16 and 25 indicates moderate anxiety, and between 26 and 63 indicates severe anxiety.

SECONDARY OUTCOMES:
Collection of post-training data | two month
  Mothers will be given breastfeeding training 3 times with a simple explanation method. The first simple explanation is breastfeeding education in the 2nd-5th postpartum period. Between days, second simple explanation breastfeeding education postpartum13th-17th. Between days, the third simple explanation breastfeeding education is between 30th and 42nd postpartum. will be given between days. The Breastfeeding Self-Efficacy Scale will be administered after each breastfeeding training.
  The Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert-type scale consisting of 14 items (1: not at all confident and 5: always confident). The lowest score that can be obtained from the scale is 14 and the highest score is 70. A high score indicates high breastfeeding self-efficacy.
Collection of post-training data | two month
  Beck Anxiety Scale will be applied after each breastfeeding education given with a simple explanation method.
  The scale, consisting of 21 questions, is a 4-point Likert type. Each item in the scale is scored between 0 (not at all) and 3 (serious). The lowest score that can be obtained from the scale is 0 and the highest score is 63. An increase in the score obtained from the scale indicates that the individual's anxiety increases. A total score from the scale between 8 and 15 indicates mild anxiety, between 16 and 25 indicates moderate anxiety, and between 26 and 63 indicates severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: gülhan akdemir, Study Director — Igdir University
Locations (1):
- Dr. Nevruz Erez State Hospital, Iğdır, Turkey (Türkiye)